CLINICAL TRIAL: NCT03775226
Title: An Early Feasibility Study to Assess Safety and Efficacy of the ChampioNIR® SFA Stent in the Treatment of Patients With Femoro-Popliteal Disease
Brief Title: ChampioNIR® SFA Stent EFS Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study objective was achieved. Patients are no longer being examined or receiving intervention.
Sponsor: Medinol Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SFA-Israel-001
Record Dates: First submitted 2018-11-21; First posted 2018-12-13 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single are (Experimental): This study is designed as an early feasibility, prospective, open label, single arm study. 30 patients with infra-inguinal peripheral arterial disease appropriate for treatment with a femoro-popliteal stent will be treated with ChampioNIR® SFA stent implantation.
  Interventions: Device: ChampioNIR® SFA Stent

INTERVENTIONS:
Device: ChampioNIR® SFA Stent — The ChampioNIR® SFA Stent is composed of a Nitinol alloy structure with an elastomeric micro-fiber mesh and is designed specifically to be used in the peripheral vasculature. The stent is characterized by high flexibility, strong radial support and high resistance to fractures, as well as high deliverability and precise positioning.
  Other Names: ChampioNIR®

SUMMARY:
An Early Feasibility Study to Assess Safety and Efficacy of the ChampioNIR® SFA Stent in the Treatment of Patients with Femoro-Popliteal Disease

DETAILED DESCRIPTION:
Device Overview:

The ChampioNIR® SFA Stent is composed of a Nitinol alloy structure with an elastomeric micro-fiber mesh and is designed specifically to be used in the peripheral vasculature. The stent is characterized by high flexibility, strong radial support and high resistance to fractures, as well as high deliverability and precise positioning.

Objectives:

* To assess the safety and feasibility of delivery and implantation of ChampioNIR® SFA Stent.
* To assess the early and long term ability of the stent to maintain vessel patency.
* To assess the long term safety of the ChampioNIR® SFA Stent.

This study is designed as an early feasibility, prospective, open label, single arm study. 30 patients with infra-inguinal peripheral arterial disease appropriate for treatment with a femoro-popliteal stent will be treated with ChampioNIR® SFA stent implantation. All enrolled patients will be followed up at 30 days and up to 36 months. The follow-up visits will include patency evaluation by duplex ultrasound.

Primary efficacy endpoint: Primary patency of the target lesion at 6 months. Primary patency is defined as the absence of target lesion restenosis (defined by Duplex ultrasound (US) peak systolic velocity ratio (PSVR) >2.4) Primary safety endpoint: Composite rate of freedom from all-cause death, target vessel revascularization or any amputation of the index limb through 30 days following stent implantation.

Secondary efficacy endpoints:

1. Primary patency defined by Duplex US peak systolic velocity ratio (absence of restenosis which defined by Duplex US PSVR >2.4) at 30 days and 12 months.
2. Acute device success, defined as achievement of a final residual diameter stenosis of <50% by Quantitative Angiography (QA), using the assigned treatment only.
3. Acute procedural success, defined as device success with <50% residual stenosis immediately after stent placement or mean trans-stenotic pressure gradient <5 mmHg, and without the occurrence of death, amputation or repeat revascularization of the target lesion during the hospital stay.
4. Acute technical success, defined as the attainment of <50% residual stenosis by QA by any percutaneous method as determined by the angiographic core laboratory.
5. The following endpoints at 30 days 6, 12, 24 and 36 months:

   * Secondary Patency (absence of restenosis which is defined as Duplex US PSVR ≥ 2.4)
   * Change of Rutherford classification from baseline
   * Change of resting ankle-brachial index (ABI) from baseline
   * Change in walking impairment questionnaire from baseline
   * Change in six minute walk test from baseline

Secondary safety endpoints:

1. Combined rate of death at 30 days, target lesion revascularization (TVR), index limb amputation and increase in Rutherford-Becker Classification by ≥2 classes (as compared to post-procedural assessment) throughout 12 months.
2. Stent fracture at 30 days 6, 12, 24 and 36 months. Stent fractures will be analyzed by a two-view X-ray evaluation by a designated core laboratory, compared with a baseline two-view X-ray taken before discharge and defined as type I, II, III, IV or V as follows:

   * Type I - a single strut fracture only.
   * Type II - multiple single nitinol stent fractures that can occur at different sites.
   * Type III - multiple nitinol stent fractures resulting in complete transverse linear fracture but without stent displacement.
   * Type IV - a complete transverse linear type III fracture with stent displacement.
   * Type V - a spiral dissection of a stent.
3. Freedom at 30 days from all-cause death, index limb amputation above the ankle and TVR.
4. The following endpoints will be assessed at 30 days, 6, 12, 24 and 36 months:

   1. All-cause death
   2. Amputation (above the ankle)-Free Survival (AFS)
   3. Target Vessel Revascularization (TVR)
   4. Re-intervention for treatment of thrombosis of the target vessel or embolization to its distal vasculature
5. Major Adverse Limb Events (MALE) at 30 days, 6, 12, 24 and 36 months:

   1. Stent thrombosis
   2. Clinically apparent distal embolization (defined as causing end-organ damage, e.g. lower extremity ulceration, tissue necrosis, or gangrene)
   3. Procedure-related arterial rupture
   4. Acute limb ischemia
   5. Target limb amputation
   6. Procedure related bleeding event requiring transfusion

Sample Size and Statistical Analysis:

The study is an early feasibility study and is not powered towards finding significant differences in the primary endpoints. The sample size of up to 30 patients will allow for the evaluation of feasibility and safety of the procedure, to support the initiation of a pivotal study. No formal statistical power calculations were conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and of age of legal consent.
2. Subject has lifestyle limiting claudication or rest pain (Rutherford-Becker scale 2-4) with a resting ankle-brachial index/toe-brachial index (ABI/TBI) <0.90/0.80.
3. A single superficial femoral artery lesion with >50% stenosis or total occlusion.
4. Stenotic lesion(s) or occluded length within the same vessel (one long or multiple serial lesions) ≥ 40 mm to ≤ 140 mm.
5. Reference vessel diameter (RVD) ≥ 3.0 mm and ≤ 6.0 mm by visual assessment.
6. Target lesion located with the distal point at least 3 cm above the knee joint, defined as the distal end of the femur at the knee joint, and proximal point at least 2 cm below the origin of the profunda femoris (deep femoral artery).
7. Patent infra-popliteal and popliteal artery, i.e., single vessel runoff or better with at least one of three vessels patent (<50% stenosis) to the ankle or foot.
8. The target lesion(s) can be successfully crossed with a guide wire and dilated.
9. The subject is eligible for standard surgical repair, if necessary.
10. Subjects are willing to comply with scheduled visits and tests and are able and willing to provide informed consent.

Exclusion Criteria:

1. Thrombophlebitis or deep venous thrombus, within the previous 30 days.
2. Presence of thrombus in the treated vessel as visualized by angiography, prior to crossing the lesion.
3. Thrombolysis of the target vessel within 72 hours prior to the index procedure, where complete resolution of the thrombus was not achieved.
4. Poor aortoiliac or common femoral "inflow" (i.e. angiographically defined >50% stenosis of the iliac or common femoral artery) that would be deemed inadequate to support a femoro-popliteal bypass graft and was not successfully treated prior to treatment of the target lesion.
5. Presence of residual ≥30% stenosis after either PTA or stenting of the inflow lesion.
6. Presence of an ipsilateral arterial artificial graft.
7. Ipsilateral femoral aneurysm or aneurysm in the SFA or popliteal artery.
8. Lesions in contralateral SFA/PPA that require intervention during the index procedure, or within 30 days before or after the index procedure;
9. Required stent placement (in the target or any other lesion) via a retrograde approach.
10. Required stent placement (in the target or any other lesion) across or within 0.5 cm of the SFA / PFA bifurcation.
11. Procedures which are pre-determined to require stent-in-stent placement to obtain patency, such as in-stent restenosis.
12. Significant vessel tortuosity or other parameters prohibiting access to the lesion or 90° tortuosity which would prevent delivery of the stent device.
13. Required stent placement within 1 cm of a previously (in a former procedure) deployed stent.
14. Use of atherectomy or other atheroablative (e.g. cryoplasty) devices at the time of index procedure.
15. Restenotic lesion that had previously been treated by atherectomy, laser or cryoplasty within 3 months of the index procedure.
16. Subject has tissue loss, defined as Rutherford-Becker classification category 5 or 6.
17. Coronary intervention within 7 days prior to or planned within 30 days after the treatment of the target lesion.
18. Stroke within the previous 90 days.
19. Known allergies to any of the following: aspirin, P2Y12 inhibitors (clopidogrel bisulfate, prasugrel, OR ticagrelor), heparin OR bivalirudin, nitinol (nickel titanium), or contrast agent, that cannot be medically managed.
20. Receiving dialysis or immunosuppressant therapy within the previous 30 days.
21. Known or suspected active infection at the time of the procedure.
22. History of neutropenia, coagulopathy, or thrombocytopenia.
23. Known bleeding or hypercoagulability disorder or significant anemia (Hb<8.0) that cannot be corrected.
24. Platelet count <80,000/μL
25. International normalized ratio (INR) > 1.5
26. GFR <30 ml/min by Cockroft-Gault.
27. Subject requires general anesthesia for the procedure.
28. Subject has a co-morbid illness that may result in a life expectancy of less than 1 year
29. Planned use of a drug coated balloon (DCB) during the index procedure.
30. Pregnant women or women of child bearing potential who do not have a negative serum or urine pregnancy test documented within 7 days prior to enrollment;
31. Subject is participating in any investigational study that has not yet reached its primary endpoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-10-27 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Primary patency of the target lesion at 6 months. | 6 months
  Primary patency is defined as the absence of target lesion restenosis (defined by Duplex ultrasound (US) peak systolic velocity ratio (PSVR) >2.4)
Composite rate of freedom | 30 Day
  from all-cause death, target vessel revascularization or any amputation of the index limb through 30 days following stent implantation.

SECONDARY OUTCOMES:
Primary patency defined by Duplex US | 30 days and 12 months.
  Primary patency defined by Duplex US peak systolic velocity ratio (absence of restenosis which defined by Duplex US PSVR >2.4
Acute device success | index procedure
  defined as achievement of a final residual diameter stenosis of <50% by Quantitative Angiography (QA), using the assigned treatment only.
Acute procedural success | index procedure
  defined as device success with <50% residual stenosis immediately after stent placement or mean trans-stenotic pressure gradient <5 mmHg, and without the occurrence of death, amputation or repeat revascularization of the target lesion during the hospital stay.
Acute technical success | index procedure
  defined as the attainment of <50% residual stenosis by QA by any percutaneous method as determined by the angiographic core laboratory.
Secondary Patency absence of restenosis which is defined as Duplex US | 30 days 6, 12, 24 and 36 months
  Secondary Patency (absence of restenosis which is defined as Duplex US PSVR ≥ 2.4)
Combined rate 30 day | 12 months
  of death at 30 days, target lesion revascularization (TVR), index limb amputation and increase in Rutherford-Becker Classification by ≥2 classes (as compared to post-procedural assessment)
Stent fractures will be analyzed by a two-view X-ray evaluation by a designated core laboratory, compared with a baseline two-view X-ray taken before discharge and defined as type I, II, III, IV or V as follow | 30 days 6, 12, 24 and 36 months
  * Type I - a single strut fracture only.
  * Type II - multiple single nitinol stent fractures that can occur at different sites.
  * Type III - multiple nitinol stent fractures resulting in complete transverse linear fracture but without stent displacement.
  * Type IV - a complete transverse linear type III fracture with stent displacement.
  * Type V - a spiral dissection of a stent.
Freedom from all-cause death, index limb amputation above the ankle and TVR. | 30 days
  Clinical: The number of patients who die from all causes
All-cause death | 30 days, 6, 12, 24 and 36 months
  Clinical: The number of patients who die from all causes
The following Major Adverse Limb Events will be evaluated either by angiography or clinical examination. These will be assessed by reviewing angiograms by the core-lab and clinical events will be adjudicated by a CEC | 30 days, 6, 12, 24 and 36 months
  1. Stent thrombosis
  2. Clinically apparent distal embolization (defined as causing end-organ damage, e.g. lower extremity ulceration, tissue necrosis, or gangrene)
  3. Procedure-related arterial rupture
  4. Acute limb ischemia
  5. Target limb amputation
  6. Procedure related bleeding event requiring transfusion
  These are clinical events, the unit of measure for all is - number of patients with any event
Rutherford classification | 30 days 6, 12, 24 and 36 months
  Change of Rutherford classification from baseline
  It is defined as follows, with increasing severity:
  1. - Mild Claudication - short duration
  2. - Moderate Claudication - moderate exercise
  3. - Severe Claudication - minor exertion
  4. - Rest Pain
  5. - Minor Tissue Loss
  6. - Major Tissue Loss
resting ankle-brachial index | 30 days 6, 12, 24 and 36 months
  Change of resting ankle-brachial index (ABI) from baseline
  Ankle Brachial Index (ABI) is a standard measure defined as:
  The systolic blood pressure at the ankle divided by the systolic blood pressure at the upper arm (brachial artery) A ratio below 0.9 is considered significant
walking impairment questionnaire | 30 days 6, 12, 24 and 36 months
  Change in walking impairment questionnaire from baseline The questionnaire will be used to assess walking capability in patients with Peripheral Arterial Disease (to evaluate the walking impairment and the efficacy of an intervention to improve walking ability in patients with Peripheral Arterial Disease, PAD).\ The patients will be required to address their walking difficulties and grade them on an increased severity scale.
six minute walk test | 30 days 6, 12, 24 and 36 months
  Change in six minute walk test from baseline
Amputation (above the ankle) | 30 days, 6, 12, 24 and 36 months
  Amputation (above the ankle)-Free Survival (AFS)
Target Vessel Revascularization | 30 days, 6, 12, 24 and 36 months
  Target Vessel Revascularization (TVR) Will be measured by the number of patients with the event
Re-intervention for treatment of thrombosis of the target vessel or embolization to its distal vasculature | 30 days, 6, 12, 24 and 36 months
  Re-intervention for treatment of thrombosis of the target vessel or embolization to its distal vasculature Will be measured by the number of patients with the event

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: Undecided